CLINICAL TRIAL: NCT01691495
Title: ARIXTRA® Physician Adherence to the Prescribing Information in Isolated Superficial Vein Thrombosis (SVT) Patients.
Brief Title: ARIXTRA® Adherence in SVT Patients.
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115280
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Thrombosis, Venous
Keywords: Physician Adherence; superficial vein thrombosis; Fondaparinux
MeSH Terms: conditions — Venous Thrombosis | interventions — Fondaparinux

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Superficial Vein Thrombosis (SVT): A representative of geographical regions of patients with Superficial Vein Thrombosis (SVT) who live in several EU countries.
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux — Physician adherence study to Fondaparinux prescribing information for patients with Superficial Vein Thrombosis (SVT) of the lower limbs

SUMMARY:
Fondaparinux is an anticoagulant used in the prevention and treatment of thromboembolic disease. It has recently been approved in the European Union (EU) for the treatment of patients with isolated superficial vein thrombosis (SVT), i.e. without concomitant deep vein thrombosis (DVT), of the lower limbs. As part of EU approval, GlaxoSmithKline (GSK) committed to evaluate physicians' adherence to fondaparinux prescribing information regarding proper diagnosis and dosing for the treatment of SVT.

The primary objective is to evaluate physicians' adherence to fondaparinux prescribing information for the treatment of patients with SVT without concomitant DVT.

The study is designed as a non-interventional, retrospective chart review of patients prescribed fondaparinux to treat their SVT. The study will be conducted in several EU countries.

ARIXTRA® is a registered trademark of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SVT
* Prescribed fondaparinux for the treatment of SVT
* Age 18 years or older

Exclusion Criteria:

* Patients should not have been involved in any clinical trial that could influence SVT treatment during the observational period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 12 clinical sites representative of geographical regions of several EU countries, targeting physician adherence to prescribing in approximately 840 patients with SVT.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be a measure of physician adherence. | 2
  adherence described as the percentage of patients for whom both an ultrasound (or other objective measure) was performed in order to rule out concomitant DVT prior to patients commencing fondaparinux

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline